CLINICAL TRIAL: NCT03444415
Title: Effectiveness of a Motivational Interviewing-based Intervention From Pregnancy to 2 Years Old.
Brief Title: Effectiveness of a Motivational Interviewing-based Intervention From Pregnancy to 2 Years of Age.
Acronym: PROGESPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROGESPI
Record Dates: First submitted 2017-12-12; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2017-12

CONDITIONS: Childhood Obesity Prevention
Keywords: Obesity; Children; Pregnancy; Motivational interview; Family Care; Primary Care
MeSH Terms: conditions — Obesity | interventions — Motivational Interviewing; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing in groups (Experimental): The Intervention is performed at Primary Care Centers by health professionals (General Practitioners, Nurses, Pediatricians and Midwives), during pregnancy and the first 2 years of the child. Researchers will be trained in motivational interviewing and group dynamics. Intervention consists of six 90 minutes workshops, two of those during pregnancy and the other four within the following two years after the birth of the children. They intend to encourage the shift towards healthy lifestyles to parents on issues related to diet, physical activity and smoking habit, encourage breastfeeding and increase their knowledge and self-efficacy to promote healthy habits regarding diet, physical activity and sleep habits of their children.
  Interventions: Other: Motivational interviewing in groups
- Control Group (Other): Control Group: Usual Care as established in the "Programa Integral de Atención a la Mujer" (Comprehensive Program of Woman Assistance) and the "Programa de Atención al Niño Sano" (Well Child Program) in the Servicio Murciano de Salud.
  Parents will receive information about height, weight, and BMI percentile provided by a health professional during usual well child visits.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Motivational interviewing in groups — Intervention consists of six 90 minutes workshops, two of those during pregnancy and the other four within the following two years after the birth of the children.
  Arms: Motivational interviewing in groups
Other: Usual care — Parents will receive information about height, weight, and BMI percentile provided by a health professional during usual well child visits
  Arms: Control Group

SUMMARY:
The main objective of this study is to evaluate the effect of an early and intensive intervention, based on techniques of effective counseling on healthy habits for parents, in order to reduce mean BMI at 2 years of age Secondly, the investigators will analyze the weighted increase of children's BMI, the eating habits of parents and children, duration of breastfeeding, physical activity level of parents and children and the children sleeping habits. In order to achieve it, the investigators have developed a randomized trial by Primary Care Centers, controlled by two parallel groups of study, open and multicenter study. The investigator team will recruit 414 pregnant women bwtween 12 and 16 weeks of gestation who will or will not receive an intervention, depending on their Primary Care Centers. The investigators will develop an intervention for parents, based on effective counseling techniques which are grounded on Motivational Interviewing approach with the objective of transmitting habits to reach a healthy lifestyle. The intervention consists in six workshops (90 minutes long), two prenatal and four postnatal, directed by professionals of the Field Researchers Basic Group (Family Practitioners, Pediatricians, Nurses and Midwives). Previously the field researchers will receive specialized training. This intervention will be compared to the usual model of care for children and women.

ELIGIBILITY:
Inclusion Criteria:

Will be included all pregnant women who have given their consent and who meet the following inclusion criteria:

* Attended in Primary Care Centers and not planning to change their place of residence in the period covered by the study.
* Women over 18 years of age.
* Gestational age between 12 and 16 weeks.
* Women whose pregnancy is liable of follow-up in Primary Care.

Exclusion Criteria:

* Women who cannot communicate in Spanish.
* Women with metabolic diseases that modify their weight (diabetes, hypothyroidism, hyperthyroidism, etc.).
* Maternal history of a serious medical or psychiatric illness or drug or alcohol abuse.
* Multiple pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 414 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
BMI | 2 years of age
  The investigator team will collect weight and height, calculate the BMI and we will work out the BMI Z-score according to WHO growth standards.

SECONDARY OUTCOMES:
Weight growth rate | 2 years of age
  WHO standardS
Food intake habits in parents | 2 years of age
  PREDIMED study questionnaire
Physical activity in parents: | 2 years of age
  International Physical Activity Questionnaire (IPAQ)
Smoking habit in parents (self-reported): measuring the percentage of parents who smoke, consumption of cigarettes per day, and their level of motivation to quit smoking through the Richmond Test. | 2 years of age
  Richmond Test.
Anthropometry of parents: | 2 years of age
  Weight and height will be combined to report BMI in kg/m^2
Duration of breastfeeding | 2 years of age
  The investigator team will measure the time of exclusive and mixed breastfeeding, in months, according to the regarding questions of the National Health Survey 2011-2012.
Children's dietary habits | 2 years of age
  PREDIMED study questionnaire
Physical Activity patterns in children | 2 years of age
  PREDIMED study questionnaire
Sleep habits | 2 years of age
  PREDIMED study questionnaire
Socio - demographic variables: Number of siblings, country of origin, educational level and social class, according to the proposal of the Spanish Society of Epidemiology and the Spanish Society of Family and Community Medicine. | 2 years of age
  PREDIMED study questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Pérez López, Principal Investigator — SMS
Locations (1):
- Pedro Pérez López, Murcia, Alcantarilla-Sangonera, Spain

IPD SHARING:
Plan to Share IPD: Undecided